CLINICAL TRIAL: NCT04638855
Title: A Placebo Comparative, Evaluator Blinded, Randomized, Multi-center Study to Evaluate the Efficacy and Safety of Medicurtain® in Patients With Hysteroscopy
Brief Title: The Efficacy and Safety of Medicurtain® in Patients With Hysteroscopy (Pivotal Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UMT2009-SP-ASMC-0401
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Intrauterine Synechiae; Tissue Adhesion, Surgery-Induced
Keywords: Medicurtain; Sodium hyaluronate; Anti-adhesion barrier
MeSH Terms: conditions — Gynatresia; Tissue Adhesions

STUDY DESIGN:
Intervention Model Description: Pivotal study (Determine effectiveness and adverse effects)
Who Masked: Outcomes Assessor
Masking Description: Evaluator-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medicurtain® (Experimental): Treat Medicurtain 5ml prefilled syringe after hysteroscopy surgery
  Interventions: Device: Medicurtain®
- Placebo (Sham Comparator): No device after hysteroscopy surgery
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Medicurtain® — Anti-adhesion barrier (Medicurtain® 5ml prefilled syringe after hysteroscopy surgery)
  Arms: Medicurtain®
Device: Placebo — No device after hysteroscopy surgery
  Arms: Placebo

SUMMARY:
This study was designed to assess the safety and efficacy of MEDICURTAIN, an adhesion barrier in patients who underwent hysteroscopy with uterine polyp or endometrial myoma or missed abortion (uterine lesion suspected to be associated with pregnancy) or intrauterine adhesion. Adhesion formation in both groups was evaluated by the grading scale and photographs taken during the follow up to evaluate the safety and efficacy of the product.

DETAILED DESCRIPTION:
This study was designed as a multi-center, randomized, evaluator-blinded and placebo-comparative study. A woman aged 20-80 years scheduled for the hysteroscopy was eligible to participate in the study. Subject screening was conducted for the subject who signed an informed consent form. Subjects who met the inclusion/exclusion criteria were randomly assigned into either treatment or no-treatment control group. Follow-up visits were performed at 1 week (Visit 2) and 4 weeks (Visit 3) after the index surgery. Telephone call is made between 1 to 2 weeks prior to the Visit 3 for the information for the follow-up visit and check-up.

At Visit 2 (at Week 1 after the index surgery, a window of ± 2 days was allowed), assessments to identify adverse events and general health conditions, and surgery satisfaction survey were performed. At Visit 3 (at Week 4 ± 4 days), adverse event assessments and general satisfaction survey were performed, and adhesion formations and grades were evaluated. The presence or absence of adhesions, and their grades at Visit 3 (at Week 4 ± 4 days) were assessed in an evaluator-independent manner.

Adhesion formations rate (Primary endpoint) and adhesion grade(secondary endpoint) were assessed at Week 4 after the index surgery (Visit 3), based on the video clips and still images captured via a video monitor during a second-look hysteroscopy, by inserting the hysteroscope (5 -10 mm diameter) into the uterine through the vagina; and graded in an evaluator-blinded manner by an independent evaluator, who did not take part in the index surgery or application of Medicurtain®. Intrauterine adhesion grades were assessed by using the American Fertility Society (AFS) adhesion score established in 1988. It was classified as 4 grading scales (0, 1, 2 and 3 grade). Grade 0 (none) means no adhesion, while Grade 1 to Grade 3 means there are adhesions and severity increased with the grade. Adhesion formation rate and grade in the treated or in the non-treated control groups were compared and evaluated using the Grade 0 to 3 adhesion scoring system.

ELIGIBILITY:
Inclusion Criteria:

1. Woman who is between 20~80 years of age.
2. Woman who is reserved elective hysteroscopy for

   * Uterine polyp
   * Uterine (endometrium) myoma
   * Missed miscarriage (uterine lesion suspected to be associated with pregnancy)
   * Adhesion in uterine
3. Woman who signed an informed consent form prior to the investigation.

Exclusion Criteria:

1. Presence of tumor or inflammatory disease in other organs.
2. Subject who is not eligible for anesthesia or re-operation due to other disease confirmed by investigator.
3. Subject who is not eligible for re-operation or hysteroscopy
4. Any condition which made a subject unsuitable for inclusion in the discretion of the Investigator will be excluded.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 223 (Actual)
Dates: Start 2010-09-08 (Actual); Primary Completion 2011-12-03 (Actual); Study Completion 2011-12-03 (Actual)

PRIMARY OUTCOMES:
Outcome Measure: comparison between treated group and untreated control group for the adhesion rate | 4 weeks
  Adhesion rate: {(number of subjects occurred adhesion formation for each group)/ (number of subjects for each group)} * 100

SECONDARY OUTCOMES:
Comparison of Adhesion Grade between treated group and untreated control group | 4 weeks
  Adhesive grade evaluation standards are classified into Grade 0(Non), Grade 1(Mild), Grade 2(Moderate), Grade 3(Severe).
The incidence rate of adverse events | follow up to 4 weeks
  Safety and tolerability by collecting adverse events (AEs)
The incidence rate of adverse drug reaction | follow up to 4 weeks
  Safety and tolerability by collecting adverse drug reaction (ADRs)
The incidence rate of serious adverse events | follow up to 4 weeks
  Safety and tolerability by collecting serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Byeongseok Lee, MD, Principal Investigator — Gangnam Severance Hospital, 712 Eonju-ro, Gangnam, Seoul, South Korea; Youngsik Choi, MD, Principal Investigator — Severance Hospital, 134 Sinchon-dong, Seodaemun-gu, Seoul, South Korea; Sun Hee Cha, MD, Principal Investigator — Bundang CHA Medical Center, 351 Yatap-dong, Seongnam-si, Gyeonggi-do, South Korea; Joomyung Kim, MD, Principal Investigator — CHEIL General Hospital & Women's Healthcare Center, 1-19 Mukjeong-dong, Jung-gu, Seoul, South Korea; Ki-Hwan Lee, MD, Principal Investigator — Chungnam National University Hospital, 33 Munhwa-ro, Jung-gu, Daejeon, South Korea; In Taek Hwang, MD, Principal Investigator — Daejeon Eulji Medical Center, Dunsan-2-dong, Seo-gu, Daejeon, South Korea
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No